CLINICAL TRIAL: NCT06708481
Title: Clinical Outcome of Resin Infiltration Vs Self-Assembling Peptide (P11-4) in Treating White Spot Lesion - a Randomized Clinical Trial
Brief Title: Resin Infiltration Vs Self-Assembling Peptide (P11-4) in Treating White Spot Lesions
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: October 6 University (Other)
Collaborators: Al-Azhar University (Other); University of Science and Technology of Fujairah (Unknown)
Responsible Party: Principal Investigator, Dina El Kharadly, Lecturer in Pediatric Dentistry Department, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P-PD-24-03
Record Dates: First submitted 2024-08-28; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: White Spot Lesion
Keywords: Resin Infilteration , white spot lesions , Self assembling peptide, remineralization
MeSH Terms: interventions — icon infiltrant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Self-Assembling Peptide (P11-4) (Experimental): self-assembling peptide in a brush-on liquid applied after cleaning and chemical preparation.The P11-4 peptide, called Curodont Repair (Credentis; now manufactured by vVARDIS)
  Interventions: Drug: P11-4, a self-assembling peptide
- Self-Assembling Peptide (P11-4) with fluoride varnish (Experimental): CR Fluoride Plus (CRFP) (Credentis; now manufactured by vVARDIS) also includes 500 ppm sodium fluoride and is registered with the US Food and Drug Administration (NDC 72247-101) as an anticaries drug under the fluoride monograph (21CFR355).
  Interventions: Drug: P11-4, a self-assembling peptide with flouride
- Resin Infilteration (Active Comparator): ICON® contains 15% HCl as an etchant, ethanol as a dehydrating agent, and triethylene glycol dimethacrylate (TEGDMA) resin as an infiltrant
  Interventions: Drug: resin infilteration

INTERVENTIONS:
Drug: P11-4, a self-assembling peptide — rationally designed peptide, the monomers of which self-assemble into a biocompatible fibrillar scaffold that mimics the enamel matrix in response to particular environmental cues
  Other Names: Curodont- repair
  Arms: Self-Assembling Peptide (P11-4)
Drug: P11-4, a self-assembling peptide with flouride — self assembling peptide with 500 ppm sodium fluoride
  Other Names: Curodont- repair with fouride
  Arms: Self-Assembling Peptide (P11-4) with fluoride varnish
Drug: resin infilteration — Improvement of white spot lesions appearance by infiltration occurs due to a change in the refractive index since the refractive index of enamel (1.62-1.65) is different than that of air (1.00). Infiltration of the lesions with an infiltrate that has a refractive index of 1.52 is able to mask the lesion
  Other Names: Icon
  Arms: Resin Infilteration

SUMMARY:
Clinical assessment of the effectiveness of two treatment modalities (self-assembling peptide (P11-4) (alone or combined with fluoride) and resin infiltration) for treating white spot lesions

DETAILED DESCRIPTION:
Patient/population:

Patients that range from 7-14 years of age with with at least one non-cavitated WSL located on smooth surfaces of maxillary or mandibular permanent teeth and comparable in size, opacity, and whitish appearance.

Intervention:

I1: Self-Assembling Peptide (P11-4) I2: Self-Assembling Peptide (P11-4) with fluoride varnish

Comparator Resin Infiltration

Outcome:

Primary outcome

* Esthetic Improvement of white spot lesion

Outcome measure: Photographic analysis Outcome measuring Device: Image analysis to calculate change in area ratio of WSL to the labial surface using Photoshop software.

Outcome measuring unit: change in Percentage

• Tooth remineralization

1. Outcome measure: International Caries Detection and Assessment System (ICDAS) score.

   Outcome measuring Device: Visual and Clinical examination by operator Outcome measuring Unit : Numerical score from 0-6
2. Outcome measure: Quantitative light Fluorescence score from WSL Outcome measuring Device: Diagnodent Pen Outcome measuring Unit: Numerical score from 0-99

Secondary outcome

Outcome measure: Patient Satisfaction Outcome measuring Device Likert 5-point faces scale ranging from very sad to very happy

Outcome measuring Unit :Numerical score from 1-5

Study design: Randomized clinical trial Time: 6 months

ELIGIBILITY:
Inclusion Criteria:

* Age (a range from 7-14 years of age was determined)
* Good general health (absence of disease/no handicaps, to ensure oral care at home)
* Preserved pulp vitality of the teeth.
* Consolidated oral care daily.
* Agreement by patient and parents (or guardians) to participate in the study

Exclusion Criteria:

* Patients with periodontal diseases (periodontal pockets or dental mobility) or radiologically identified pathologies (periapical radiolucency).
* Teeth revealing any restorations were excluded from the current study.
* Any previous or planned WSL treatment.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Esthetic Improvement of white spot lesion | 6 months
  Outcome Measure:
  Photographic analysis
  Outcome measuring device:
  Image analysis to calculate change in area ratio of WSL to the labial surface using Photoshop software
  Outcome measuring unit:
  Percentage change
Tooth remineralization | 6 months
  ICDAS score
  Outcome Measure:
  ICDAS score
  Outcome measuring device:
  Visual and Clinical examination by operator
  Outcome measuring unit:
  Numerical value from 0-6
  Outcome Measure:
  Quantitative Light Fluorescence score from WSL
  Outcome measuring device:
  Diagnodent pen
  Outcome measuring unit:
  Numerical value ranging from 0 to 99

SECONDARY OUTCOMES:
Patient Satisfaction | 6 months
  Likert 5-point faces scale ranging from very sad to very happy

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University, Cairo, Giza Governorate, Egypt